CLINICAL TRIAL: NCT00964262
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Dose-escalating Study to Evaluate Safety and Pharmacokinetics/Pharmacodynamics of SR Exenatide (PT302) After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: A Study to Evaluate Safety and Pharmacokinetics/Pharmacodynamics of Sustained Release(SR) Exenatide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PepE01
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; SR exenatide; Peptron
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SR Exenatide (PT302) (Experimental): Intervention: Drug: SR Exenatide (PT302)
  Interventions: Drug: SR Exenatide (PT302); Drug: Placebo

INTERVENTIONS:
Drug: SR Exenatide (PT302) — 0.5 mg, 1.0 mg, 2.0 mg and 4.0 mg dosage(dose escalation), single subcutaneous injection
Drug: Placebo — Plcacebo of each doasage, single subcutanoeus injection

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and pharmacodynamics of SR exenatide (PT302) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20-45 years at screening
* Body weight over 50 kg, inclusive, and within 20% of ideal body weight

Exclusion Criteria:

* Has a present illness or medical history of hepatic, renal, respiratory, cardiovascular disease, blood tumor, mental disorder, and endocrinologic disorder, especially diabetes mellitus
* Has a sign or symptom or history related to an acute or chronic pancreatitis
* Has a known allergy or hypersensitivity to exenatide or other drugs such as aspirin, antibiotics, and so on
* Has ever been exposed to exenatide
* Shows SBP >= 150 mmHg or <= 90 mmHg or DBP >= 100 mmHg or <= 50 mmHg
* Has a presence or history of drug abuse
* Uses any prescription drug, herbal medicine within 2 weeks or OTC drugs or vitamin within 1 week prior to study drug administration
* Has been participated in other clinical trial within 2 months
* Has experience of a blood donation during 2 months or a blood transfusion during 1 month prior to study drug administration
* Heavy smoker more than 10 cigarettes/day within 3 months prior to screening
* Continuous drinker (over 21 units/week, 1 unit = 10 g of pure alcohol) or subject who can't quit drinking nor smoking during clinical trial period
* Subjects not eligible at the discretion of investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and pharmacokinetics of SR exenatide (PT302) in healthy subjects after a single subcutaneous injection | 8 weeks

SECONDARY OUTCOMES:
To examine the effect on glucose control and pharmacodynamic parameters of SR exenatide (PT302) in healthy subjects after a single subcutaneous injection | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Gu N, Cho SH, Kim J, Shin D, Seol E, Lee H, Lim KS, Shin SG, Jang IJ, Yu KS. Pharmacokinetic properties and effects of PT302 after repeated oral glucose loading tests in a dose-escalating study. Clin Ther. 2014 Jan 1;36(1):101-14. doi: 10.1016/j.clinthera.2013.12.002. Epub 2013 Dec 27. PMID 24373998